CLINICAL TRIAL: NCT00686465
Title: Positron Emission Tomography/Computed Tomography (PET/CT) for the Diagnosis of Recurrent Cancer: a Feasibility Study. PET in Recurrent Cancer(PETREC)
Brief Title: Positron Emission Tomography/Computed Tomography (PET/CT) for the Diagnosis of Recurrent Cancer: a Feasibility Study
Acronym: PETREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2007-PETREC
Record Dates: First submitted 2008-05-22; First posted 2008-05-29 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Non-small Cell Lung Cancer; Breast Cancer; Head and Neck Cancer; Ovarian Cancer; Esophageal Cancer; Lymphoma
Keywords: recurrent cancer; PET/CT; FDG; planned management; actual treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Head and Neck Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET/CT scan (Other): PET/CT scan
  Interventions: Other: PET/CT scan

INTERVENTIONS:
Other: PET/CT scan — Patients will undergo whole body FDG-PET/CT imaging

SUMMARY:
Sometimes, cancer comes back after it has been successfully treated-a situation called recurrent cancer. When recurrent cancer is suspected, the standard approach to diagnosis is to perform a combination of imaging tests, such as x-rays, ultrasound, computed tomography (CT), magnetic resonance imaging (MRI), and nuclear medicine scans. Sometimes, however, after performing these tests it still may not be clear whether or not the cancer has come back.

Some studies have shown that a diagnostic imaging test called Positron Emission Tomography/Computed Tomography (PET/CT) may be helpful in the diagnosis of recurrent lung, breast, head and neck, ovarian or esophageal cancer or lymphoma. However, it is not clear if PET/CT can offer better results than standard approaches to diagnosis.

This feasibility study is needed to determine how common it is for a diagnosis of recurrent cancer to be unclear even after standard diagnostic imaging tests have been completed. If the enrollment goal is reached (~60 patients enrolled in 18 months), a larger clinical trial is being planned to determine if PET/CT is helpful in making the diagnosis of recurrent cancer in situations where standard imaging tests have not been helpful. It is also expected that the results of this feasibility study will help to define exactly which patients should be enrolled in this larger clinical trial of PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous history of non-small cell lung cancer, breast cancer, head and neck cancer (not thyroid cancer), ovarian cancer, esophageal cancer, or lymphoma (Hodgkin's or non-Hodgkin's) who have suspected recurrence on history and/or physical exam.
* Conventional imaging (e.g., X-ray, ultrasound, CT, MRI, bone scan) is non-diagnostic.

Exclusion Criteria:

* Age less than 18 years.
* Patient with established recurrence requiring staging of recurrent disease.
* Patients who, at the time of the initial evaluation, have already undergone PET/CT within 6 months prior to registration.
* Unable to lie supine for imaging with PET/CT.
* Pregnant or lactating female.
* Significant concurrent medical problems (e.g., uncontrolled diabetes, active cardiac disease, significant chronic obstructive pulmonary disease) making the patient unfit for further cancer therapy.
* Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The number of patients recruited in 18 months and the clinical characteristics of patients who are enrolled in the study | 21 months

SECONDARY OUTCOMES:
The proportion of patients in whom the diagnosis of recurrent cancer is confirmed (as determined by either histology or clinical follow-up at the 3 month visit) | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: John J You, MD MSc FRCPC, Principal Investigator — McMaster University; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG)
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario